CLINICAL TRIAL: NCT06986616
Title: Fibroids and the Risk of Miscarriage
Brief Title: Fibroids and the Risk of Miscarriage: a Prospective Observational Study in an Early Pregnancy Population
Acronym: FiRM
Status: Completed | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: KCH19-005
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Fibroid; Miscarriage in First Trimester; Miscarriage in Second Trimester
Keywords: fibroid; miscarriage
MeSH Terms: conditions — Leiomyoma; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases - fibroids: Women with fibroids
- Controls - no fibroids: Women without fibroids

SUMMARY:
The aim of this observational study is to whether fibroids increase the risk of miscarriage in women in our early pregnancy population.

We will be collecting lots of data detailing other factors, which may have an impact on overall health and on the risk of miscarriage (this includes age, weight, use of vitamins or progesterone supplements, postcode which is linked to national deprivation scoring status and employment status).

By collecting all this data, we hope to remove the effect of other factors and purely assess the effect that the fibroids have on the outcome in early pregnancy.

We will also be looking closely at whether the location, number or size of the fibroids can affect the pregnancy too and following up women at 24 weeks via phone. We will also look at other secondary outcomes such whether women with fibroids experience symptoms of pain or bleeding in the first or second trimester more so than their control counterparts. We will also look at the value of uterine volume as a surrogate marker of fibroid mapping.

Once all the data has been analysed, we will be able to assess whether fibroids lead to an increased risk of miscarriage. We hope that this information will be useful in counselling women affected by fibroids in the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* All women presenting at less than 10 weeks gestation either by last menstrual period or by transvaginal scan findings with an early intrauterine or ongoing pregnancy on scan

Exclusion Criteria:

* Women declining participation and follow up
* Women wishing to pursue termination of pregnancy
* Women who refuse transvaginal scan
* Multiple pregnancy
* Ectopic pregnancy
* Pregnancy of unknown location
* Embryonic demise
* Under 16
* Unable to understand - interpreting services will be used such as language line if required.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women attending the early pregnancy unit in our London hospital will be the target population.
Sampling Method: Non-Probability Sample
Enrollment: 436 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Miscarriage prior to 24 weeks | From enrollment to the end of data collection (data would be collected from 24 weeks)
  Miscarriage prior to 24 weeks - or delivery prior to 24 weeks

SECONDARY OUTCOMES:
Risk of miscarriage based on fibroid characteristics | From enrollment until data colelction (from 24 weeks)
  Risk of miscarriage based on volume, size and location of fibroids
Risk of miscarriage according to trimester | From enrollment to end of data collection (from 24 weeks)
  Risk of miscarriage according to trimester
Presence of symptoms of pain or bleeding and association with fibroids and trimester | From enrollment to end of data collection (from 24 weeks)
  Presence of symptoms of pain or bleeding and association with fibroids and trimester

OTHER OUTCOMES:
Uterine volume and value as a surrogate marker for fibroid mapping | From enrollment to end of data collection (from 24 weeks onwards).
  Can uterine volume be used as a surrogate marker for fibroid mapping - and does this have an association with miscarriage

CONTACTS AND LOCATIONS:
Locations (1):
- Early Pregnancy and Gynaecology Assessment Unit, King's College Hospital NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data is available for reasonable requests including study protocol and anonymised data.